CLINICAL TRIAL: NCT03657992
Title: Time Trend Analysis of Pulmonary Embolism Diagnosis With SPECT V/Q: a Single Institution Observational Study From 2011 to 2016
Brief Title: Time Trend Analysis of PE Diagnosis With SPECT V/Q: a Single Institution Observational Study
Acronym: TOMOBS
Status: Completed | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: TOMOBS (29BRC18.0017)
Record Dates: First submitted 2018-08-30; First posted 2018-09-05 (Actual); Last update posted 2018-09-05 (Actual); Status verified 2018-08

CONDITIONS: Pulmonary Embolism
MeSH Terms: conditions — Pulmonary Embolism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Following the implementation of SPECT V/Q imaging for PE diagnosis, the investigators previously conducted an observational study over the period 2011-2013 that showed the safety of a diagnostic management based on SPECT V/Q to rule out PE. However, PE prevalence was high (28%), which may seem a bit high as compared with other recent studies. The hypothesis was that the use of SPECT V/Q may be responsible for an overdiagnosis of PE, especially at the implementation phase of the test. The aim of this study was to perform a time trend analysis of the evolution over the years of PE diagnosis with SPECT V/Q.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent a SPECT V/Q scan performed for a suspected acute PE in the Nuclear Medicine Department of Brest University Hospital from April 2011 to December 2016

Exclusion Criteria:

* Patient under legal or judicial protection
* Patient opposed to the use of his medical data for research.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who underwent a SPECT V/Q scan performed for a suspected acute PE in the Nuclear Medicine Department of Brest University Hospital from April 2011 to December 2016
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2018-05-30 (Actual); Study Completion 2018-05-30 (Actual)

PRIMARY OUTCOMES:
Diagnostic conclusion of all SPECT V/Q scans performed for a suspected acute PE | April 2011 to December 2016
  positive, negative, or non-conclusive

SECONDARY OUTCOMES:
Risk of thromboembolic events (i.e. objectively confirmed pulmonary embolism or proximal deep vein thrombosis) during the 3-month follow-up period in patients left untreated based on a negative SPECT V/Q. | up to 3 Months following the date of the SPECT V/Q scan

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU de Brest, Brest, France